CLINICAL TRIAL: NCT04098016
Title: Feasibility of Delivering a Digital Behavioral Intervention to Increase Diet Quality Among Women Receiving WIC Benefits
Brief Title: Digital Intervention To Improve Diet Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00102702
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-08

CONDITIONS: Diet, Healthy; Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will receive: 1) tailored behavior change goals, 2) self-monitoring with tailored feedback, and 3) skills training.
  Interventions: Behavioral: Digital Intervention

INTERVENTIONS:
Behavioral: Digital Intervention — Participants will receive: 1) tailored behavior change goals, 2) self-monitoring with tailored feedback, 3) skills training.

SUMMARY:
This study will develop a digital intervention ("Healthy Roots") adapted from a previously tested adult digital obesity treatment intervention ("Track").

DETAILED DESCRIPTION:
Healthy Roots will focus on improving the clinical encounter between WIC clinicians and socioeconomically disadvantaged mothers, who are disproportionately impacted by obesity, during the first 6 months postpartum.

Prior to the clinical trial portion of this project, quantitative interviews (Aim 1) were held to explore how digital health tools can be use to improve the dietary patterns of mothers and caregivers during the early postpartum period. 13 individuals who receive WIC benefits from Piedmont Health Services will be asked to participate in a one-time interview with research staff.

Following quantitative interviews, the proposed trial (Aims 2 and 3) will test the feasibility of mothers receiving WIC benefits to participate in a pilot digital behavioral intervention to increase diet quality, which will deliver nutrition guidance for meeting recommendations outlined in the Dietary Guidelines for Americans using interactive self-monitoring and feedback, and tailored skills training. The investigator will also explore acceptability of participating in Healthy Roots among both mothers receiving WIC benefits and WIC clinicians who are delivering counseling. This will help determine the potential for this intervention to be implemented into the existing clinical WIC encounter.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Has a smartphone with a data plan and an email address;
* willing to receive daily text messages;
* receives WIC benefits from Piedmont Health Services (North Carolina)
* has a child that is 24 months or younger
* speaks English as primary language.

Exclusion Criteria:

* participating in another related clinical trial;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kay, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center - with Piedmont Health Services, Inc., Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is a feasibility trial. There will be no data to share.

REFERENCES:
- [Derived] Kay MC, Hammad NM, Herring SJ, Bennett GG. Using Interactive Text Messaging to Improve Diet Quality and Increase Redemption of Foods Approved by the Special Supplemental Nutrition Program for Women, Infants, and Children: Protocol for a Cohort Feasibility Study. JMIR Res Protoc. 2021 Dec 15;10(12):e32441. doi: 10.2196/32441. PMID 34914616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 54
Completed | 48
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 34
  Non-Hispanic Black | 14
  Non-Hispanic two or more races | 2
  Hispanic | 2
  Did not respond | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54
Healthy Eating Index-2015 score [Mean (Standard Deviation); unit: units on a scale] — The Healthy Eating Index (HEI) is a measure of diet quality used to assess how well a set of foods aligns with key recommendations of the Dietary Guidelines for Americans (DGA). The scores range from 0 to 100. A higher score reflects greater alignment with key dietary recommendations from the DGA.
  units on a scale | 49.7 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Intervention Engagement- Number of Text Messages Completed
Description: The average number of text messages completed over the 3-month intervention period. Text messages will be deployed three times a week throughout the 12-week intervention.
Time Frame: 3 months
Population: Only applicable to the intervention group.
Measure: Mean (Standard Deviation); unit: text messages
Arm/Group | Intervention
Number analyzed (Participants) | 54
text messages | 7.4 (4.6)

2. Secondary Outcome: Change in Healthy Eating Index Score
Description: The Healthy Eating Index (HEI) is a measure of diet quality used to assess how well a set of foods aligns with key recommendations of the Dietary Guidelines for Americans (DGA). The scores range from 0 to 100. A higher score reflects greater alignment with key dietary recommendations from the DGA.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 48
score on a scale | 0.8 (12.9)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT04098016/Prot_001.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT04098016/SAP_002.pdf
  • Informed Consent Form (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04098016/ICF_000.pdf